CLINICAL TRIAL: NCT03688282
Title: Wearable Vibration Device to Prevent Bone Loss in Postmenopausal Women--Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranova, L.L.C. (Industry)
Collaborators: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CRD-09-1105
Record Dates: First submitted 2018-09-19; First posted 2018-09-28 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2020-11

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Wearable belt (Sham Comparator): Device will be worn but not turned on for 30 minutes.
  Interventions: Device: Sham, wearing belt
- Wearable vibration belt (30) (Experimental): Device will be worn and turned on for 30 minute treatment.
  Interventions: Device: Wearable vibration belt

INTERVENTIONS:
Device: Wearable vibration belt — The device is worn, a wearable vibration belt, for a specified time. This will provide vibration starting at the hips.
  Arms: Wearable vibration belt (30)
Device: Sham, wearing belt — The device is worn, for a specified time. It will not be turned on during this period. It is only sham.
  Arms: Sham Wearable belt

SUMMARY:
The wearable vibration device aims to consistently deliver vibrations directly to the hip and spine and allowing use during many everyday activities. We propose that demonstrating higher rates of compliance and consistent delivery of optimal force, with accelerometer feedback, will provide a superior alternative to whole body vibration and is plausibly more effective at preventing bone loss in postmenopausal women than vibration platforms in the home setting.

DETAILED DESCRIPTION:
The goal of this study is to demonstrate that postmenopausal women will tolerate our device, have high rates of compliance with the study protocol, receive consistently therapeutic levels of vibration and see significant effects on bone turnover based on plasma markers of bone anabolism and catabolism.

The anticipated outcomes from serum draws are an improvement in two bone turnover markers after a 30 minute treatment with the WVD.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Last menstrual period at least one year prior and not more than eight years prior.
3. 19 years of age and older.
4. BMD T-score at or above -2.49 at the total hip and L1-L4 spine skeletal sites as measured by DXA.
5. Ambulatory (can walk or stand without an assistive device for a minimum of 30 minutes).
6. Able to understand spoken and written English.
7. Capable and willing to follow all study-related procedures.

Exclusion Criteria:

1. BMD T-score at or below -2.5 at the total hip and L1-L4 spine skeletal sites as measured by DXA.
2. A 10-year probability of hip fracture of > 3% or major fracture of > 20% based on results of DXA using the FRAX tool (see attached).
3. Weight > 300 lbs.
4. Are currently taking or have taken bisphosphonates within the past 12 months, estrogen replacement therapy, or drugs affecting bone such as tamoxifen or aromatase inhibitors within the past 6 months.
5. Active cancer or cancer treatment.
6. Any change in exercise in the past 3 months.
7. Fractures or major surgery within the past 6 months.
8. Medical Implants (excluding dental implants).
9. Diagnosed with Paget's disease, heart disease, uncontrolled hypertension, renal disease, chronic fatigue syndrome, herniated disc, severe peripheral neuropathy, severe osteoarthritis.
10. Any bleeding disorder or treatment with a blood thinning medication within the last 2 years.
11. Hip circumference is greater than 42 inches

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham & 30 Minute Treatment: Visit 1:
  Device will be worn but not turned on. Wearable vibration belt: The device is worn, a wearable vibration belt, for a specified time. This will provide vibration starting at the hips.
  Visit 2:
  Device will be worn and turned on for 30 minute treatment. Wearable vibration belt: The device is worn, a wearable vibration belt, for a specified time. This will provide vibration starting at the hips.
Period: Sham Treatment for 30 Minutes
Arm/Group | Sham & 30 Minute Treatment
Started | 18
Completed | 17
Not Completed | 1
Period: Washout (7 Days)
Arm/Group | Sham & 30 Minute Treatment
Started | 17
Completed | 17
Not Completed | 0
Period: Active Treatment for 30 Minutes
Arm/Group | Sham & 30 Minute Treatment
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Same subjects in the single arm (2 visits)
Groups:
- Sham & 30 Minute Treatment: Visit 1:
  Device will be worn but not turned on for 30 minute treatment. Wearable vibration belt: The device is worn, a wearable vibration belt, for a specified time. This will provide vibration starting at the hips.
  Visit 2:
  Device will be worn and turned on for 30 minute treatment. Wearable vibration belt: The device is worn, a wearable vibration belt, for a specified time. This will provide vibration starting at the hips.
Arm/Group | Sham & 30 Minute Treatment
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.41 (4.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Blood-based Biomarker of Bone Loss
Description: Percent change in NTX, a biomarker of bone loss activity measured in the blood. Percent change in NTX was determined from Baseline (pre-treatment) to 30-minutes post-treatment for the sham treatment and the active treatments. The difference in percent change was then compared between active and sham treatments.
Time Frame: Baseline and 30 minutes after completing the 30-minute treatment session
Population: All subjects that completed both treatment sessions
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Sham Treatment Session: Device will be worn but not turned on (does not deliver the active treatment) for 30 minute treatment session.
- Active Treatment Session: Device will be worn and turned on (delivers the active treatment) for 30 minute treatment session.
Arm/Group | Sham Treatment Session | Active Treatment Session
Number analyzed (Participants) | 17 | 17
Percent change | 8.8 (7.6) | -5.4 (8.8)
Statistical Analysis 1: Comparison: Sham Treatment Session vs Active Treatment Session; Test type: Superiority; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Study duration (2 weeks)
Description: Standard definitions for serious adverse event and adverse event were used.
Groups:
- Sham Treatment Session: Device will be worn but not turned on (does not deliver active treatment therapy) for the 30 minute treatment session.
- Active Treatment Session: Device will be worn and turned on (delivers active treatment therapy) for the 30 minute treatment session.
Arm/Group | Sham Treatment Session | Active Treatment Session
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT03688282/Prot_001.pdf